CLINICAL TRIAL: NCT03869983
Title: A Randomized, Double-Blind, 2-Period Crossover Trial to Determine the Relative Bioavailability of CE-Iohexol (Iohexol/Sulfobutylether-β-Cyclodextrin ( Captisol®)) Injection and Omnipaque™ (Iohexol) Injection in Healthy Adult Volunteers
Brief Title: Relative Bioavailability of CE-Iohexol (Captisol-enabled™ Iohexol) Injection and Omnipaque™ Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CyDex Pharmaceuticals, Inc. (Industry)
Collaborators: Ligand Pharmaceuticals (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Organization: Ligand Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CE-Iohexol Protocol -101; Study Number-1802282 (Other: Syneos Health)
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-03

CONDITIONS: Contrast-induced Nephropathy; Coronary Angiography
Keywords: Iohexol; Captisol®; cyclodextrin; radiographic; iodinated contrast medium; Omnipaque™
MeSH Terms: interventions — Iohexol; Injections

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, 2-period, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study with limited access to the randomization code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Comparator (Active Comparator): Omnipaque™ (iohexol) Injection, 755 mg/mL iohexol (350 mgI/mL)
  Interventions: Other: Omnipaque™ (iohexol) Injection
- Experimental (Experimental): CE-Iohexol Injection, 755 mg/mL iohexol (350 mgI/mL)/50 mg CAPTISOL®/mL
  Interventions: Other: CE-Iohexol

INTERVENTIONS:
Other: Omnipaque™ (iohexol) Injection — 755 mg/mL iohexol (350 mgI/mL), 80 mL infused intravenously over approximately 20 seconds
  Arms: Active Comparator
Other: CE-Iohexol — 755 mg/mL iohexol (350 mgI/mL)/50 mg CAPTISOL®/mL, 80 mL infused intravenously over approximately 20 seconds
  Arms: Experimental

SUMMARY:
This study is designed to compare the bioavailability of the test Product(CE-Iohexol Injection) and the reference product Iohexol Injection (Omnipaque™) following intravenous injection in normal healthy volunteers. The secondary objective is to assess the safety and tolerability of the treatments administered. Captisol® is present to improve stability and to potentially reduce the risk of contrast-induced acute kidney injury(CI-AKI) associated with iohexol administration.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, 2-period, crossover study. A total of 24 subjects will be enrolled in the study; subjects will be dosed as 2 groups of 12 subjects each. Additional subjects may be enrolled into the study to obtain the statistical power of 90%. Subjects will attend a screening visit within 28 days prior to Period 1, and eligible subjects will then return to the clinic on the evening prior to Day -1. On Day 1, prior to dosing, subjects will be randomized to receive either CE-Iohexol Injection or the reference product during the first treatment period and the alternate product during the second treatment period. In each period, the study drug will be administered after a fasting period ≥8 hours. Each dose of intravenous iohexol will be separated by a minimum of a 7-day washout period. The test or reference product (iohexol 350 mg Iodine/mL, 80 mL) will be infused at a high flow rate of 4 mL/second for a dose of 400 mgI/kg for 70 kg subject. The test or reference product will be administered using a power injector. Plasma samples for determination of iohexol concentrations will be obtained from arm #2 (the arm not used for dosing) at 0 (pre-dose), 30 seconds, 5, 10, 15, 20, 30 and 45 minutes, and 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after infusion start; the 30-second sample obtained at the end of infusion. Subjects will be discharged from the clinic on Day 3 following collection of the 48-hour blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential who are sexually active with a non-sterile male partner must be using a medically acceptable form of birth control for the duration of the trial and for 30 days after the last dose of study drug
* BMI within the range of 18.5-35 kg/m2, inclusive, and body weight > 45 kg
* No significant disease or abnormal laboratory values
* Normal vital signs, without any clinically significant abnormalities
* Normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction
* Nonsmokers defined as not having smoked in the past 3 months prior to dosing
* Estimated glomerular filtration rate (eGFR) of > 60 mL/min/1.73 m2

Exclusion Criteria:

* Known hypersensitivity or allergy to iohexol, CAPTISOL®, Omnipaque™ or its excipients
* Known hypersensitivity or allergy to iodine or radio-opaque dyes
* Women who are pregnant or breast feeding
* History or presence of asthma or other pulmonary disease, thyroid disease (hypo- or hyperthyroidism), hepatitis or other liver disease
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise a major system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Abnormal laboratory values which are considered clinically significant
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2)
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dose
* Use of medication other than topical products without significant systemic absorption, hormonal contraceptives and hormone replacement therapy
* Unwilling to refrain from consumption of alcohol within 48 hours prior to each dose administration and during any in-patient period.
* Positive urine drug screen, positive alcohol breath test or positive cotinine test at screening and upon check-in to the study facility
* History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit
* Illicit drug use,significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction
* A history of difficulty with donating blood or with the insertion of large-calibre catheter
* Donation of plasma (500 mL) within 7 days prior to drug administration.
* Hemoglobin < 128 g/L (males) and < 115 g/L (females) and hematocrit < 0.36 L/L (males) and < 0.32 L/L (females) at screening
* Any history of photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Iohexol Area Under the Concentration-Time Curve (AUC) [ Time Frame: At designated time points up to 48 hours per Period ] | 48 hours
  Blood samples are to be collected at designated time points for the determination of the iohexol AUC. (Time points for CE-Iohexol Injection: Pre-dose, 30 seconds, 5, 10, 15, 20, 30 and 45 minutes, and 1, 2, 3, 4, 6, 8, 12, 24 and 48 hrs post dose. Time points for Omnipaque™ (iohexol) Injection: Pre-dose, 30 seconds, 5, 10, 15, 20, 30 and 45 minutes, and 1, 2, 3, 4, 6, 8, 12, 24 and 48 hrs post dose).
Iohexol Maximum Plasma Concentration (Cmax) [ Time Frame: At designated time points up to 48 hours per Period ] | 48 hours
  Blood samples are to be collected at designated time points for the determination of the iohexol Cmax. (Time points for CE-Iohexol Injection: Pre-dose, 30 seconds, 5, 10, 15, 20, 30 and 45 minutes, and 1, 2, 3, 4, 6, 8, 12, 24 and 48 hrs post dose. Time points for Omnipaque™ (iohexol) Injection: Pre-dose, 30 seconds, 5, 10, 15, 20, 30 and 45 minutes, and 1, 2, 3, 4, 6, 8, 12, 24 and 48 hrs post dose).

SECONDARY OUTCOMES:
Severity of all Adverse Events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) [Time Frame: Day -1, 24h and 48h post dose]. | 30 days
  An adverse event is defined as any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. The severity of all adverse events will be graded according to the CTCAE version 4.0 from dosing until 30 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Keith Marschke, PhD, Study Director — Ligand Pharmaceuticals
Locations (1):
- Syneos Health Clinique, Québec, Quebec, Canada